CLINICAL TRIAL: NCT03196609
Title: Characteristics of the Intestinal Microbiota in Patients With Cancer (Catalogue-Onco)
Brief Title: Characteristics of the Intestinal Microbiota in Patients With Cancer
Acronym: Catalogue-Onco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Catalogue-Onco
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Oncology
Keywords: Intestinal microbiota, microbial genes, oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This cohort will consist of 55 patients as described below:
  * non-small cell lung cancer (NSCLC)
  * hepatocellular cancer:
  * colorectal cancer
  * breast cancer
  * prostate cancer
  * glioblastoma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohorte (Experimental): This cohort will consist of patients as described below:
  * 15 patients with non-small cell lung cancer (NSCLC)
  * 10 patients with hepatocellular cancer:
  * 10 patients with colorectal cancer
  * 10 patients with breast cancer
  * 10 patients with prostate cancer
  * 10 patients with glioblastoma
  Interventions: Biological: Collection of stool and serum samples

INTERVENTIONS:
Biological: Collection of stool and serum samples — During the inclusion visit (for the 5 cancer sites): Stool collection (1 tube RNA later + 1 tube DMQO-EDTA) +Blood sample (1 tube SST + 1 tube EDTA)
  1 month after treatment (only for non-small cell lung cancer): Stool collection (1 tube RNA later + 1 tube DMQO-EDTA) + Blood sample (1 tube SST + 1 tube EDTA)

SUMMARY:
In order to understand how the intestinal microbiota plays a role in the effectiveness of an anti-cancer treatment by an immune control point inhibitor, this study aims to constitute a catalog of microbial genes of a patient with cancer. This catalog will help to characterize the intestinal microbiota of cancer patients and to be able to use this catalog as a reference tool for screening the microbiota of patients treated with immune control point inhibitors. To produce this catalog, five types of cancer were selected: non-small cell lung cancer, colorectal cancer, hepatocellular carcinoma, breast cancer and prostate cancer.

The metagenomic analysis of a group of five different types of cancers introduces a lot of heterogeneity which is favorable to the richness of a catalog. For non-small cell lung cancer treated with immune control point inhibitors, two stool collections will be performed per patient (one stool collection before setting up an immune control point inhibitor and one collection after one month of being inhibited Of immune control point) to assess the impact of the immune control point inhibitor on the microbiota (pilot study). For this study, two stool collection tubes containing different preservative solutions will be used (one RNAlater tube and one DMSO-EDTA tube for Dimethylsulfoxide-Ethylene diamine tetraacetic acid).

In parallel, we will also collect samples of serum and plasma to evaluate, in a second step, protein markers in circulating blood.

DETAILED DESCRIPTION:
Primary objective: Develop a catalog of microbial genes dedicated to oncology (Onco catalog) by sequencing stool specimens from patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 75 years of age.
* Patients with one of the following types of cancer: non-small cell lung cancer, hepatocellular carcinoma, colorectal cancer, breast cancer, prostate cancer and glioblastoma
* Patients with informed consent to participate in the study.
* Affiliation to the social security system

Exclusion Criteria:

* For patients with hepatocellular cancer, patients infected with the human immunodeficiency virus (HIV)
* Patients who are unable to understand, read and / or sign informed consent
* Patients who can not collect / send stools for geographical, social or psychological reasons
* Patients with previous cancer in the 5 years preceding this study
* Persons benefiting from a system of protection for adults (including guardianship and curatorship)
* Pregnant or nursing women
* Patients with another synchronous tumor
* Patients with fecal transplant
* Patients with chronic inflammatory bowel disease (IBD)
* Patients having had in the 3 months preceding the collection of stool: colonoscopy, bariatric surgery, surgical removal of a segment of the small intestine (enteritomy or enterostomy), parenteral nutrition.
* Patients who had had antibiotic therapy within 1 month before stool collection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Microbial DNA | inclusion
  Bio-computer and bio-statistical analyzes will be carried out in order to constitute the gene catalog.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Georges-François Leclerc, Dijon
  - Hopital Universitaire Paul Brousse, Villejuif